CLINICAL TRIAL: NCT01007019
Title: A Dose-block Randomized, Double-blind, Placebo/Active-controlled, Single/Multiple Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety/Tolerability and PKs/PDs of YH4808 After Oral Administration in Healthy Male Subjects
Brief Title: Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of YH4808 After Oral Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: YCD142 (YH4808-101)
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Safety, tolerability and PK/PD
MeSH Terms: interventions — YH4808; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- YH4808 30mg (Experimental): 1.Single dose
  2.12 volunteers were administered YH4808 30mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808 30mg
- YH4808 50mg (Experimental): 1.Single dose
  2.12 volunteers were administered YH4808 50mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808 50mg
- YH4808 100mg (Experimental): 1.Single dose
  2.12 volunteers were administered YH4808 100mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808 100mg
- YH4808 200mg (Experimental): 1.Single dose
  2.12 volunteers were administered YH4808 200mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808 200mg
- YH4808 400mg (Experimental): 1.Single dose
  2.12 volunteers were administered YH4808 400mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808
- YH4808 100mg(repeat doses) (Experimental): 1.Repeat doses
  2.12 volunteers were administered YH4808 100mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808 100mg (repeat dose)
- YH4808 200mg(repeat doses) (Experimental): 1.Repeat doses
  2.16 volunteers were administered YH4808 200mg or active/placebo comparators.(YH4808:active:placebo=8:6:2)
  Interventions: Drug: YH4808 200mg (repeat dose)
- YH4808 400mg(repeat doses) (Experimental): 1.Repeat dose
  2.12 volunteers were administered YH4808 400mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808 400 mg (repeat doses)
- YH4808 600mg (Experimental): 1.Single dose
  2.12 volunteers were administered YH4808 600mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808 600mg
- YH4808 800mg (Experimental): 1.Single dose
  2.12 volunteers were administered YH4808 800mg or active/placebo comparators.(YH4808:active:placebo=8:2:2)
  Interventions: Drug: YH4808 800mg (single dose)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Esomeprazole 40mg (Active Comparator)
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: YH4808 30mg — YH4808 30mg (single dose)
  Other Names: YH4808 30mg (single dose)
  Arms: YH4808 30mg
Drug: YH4808 50mg — YH4808 50mg (single dose)
  Other Names: YH4808 50mg (single dose)
  Arms: YH4808 50mg
Drug: YH4808 100mg — YH4808 100mg (single dose)
  Other Names: YH4808 100mg (single dose)
  Arms: YH4808 100mg
Drug: YH4808 200mg — YH4808 200mg (single dose)
  Other Names: YH4808 200mg (single dose)
  Arms: YH4808 200mg
Drug: YH4808 — YH4808 400mg (single dose)
  Other Names: YH4808 400mg (single dose)
  Arms: YH4808 400mg
Drug: YH4808 100mg (repeat dose) — YH4808 100mg (repeat dose)
  Arms: YH4808 100mg(repeat doses)
Drug: YH4808 200mg (repeat dose) — YH4808 200mg (repeat dose)
  Arms: YH4808 200mg(repeat doses)
Drug: YH4808 600mg — YH4808 600mg
  Arms: YH4808 600mg
Drug: YH4808 800mg (single dose) — YH4808 800mg (single dose)
  Arms: YH4808 800mg
Drug: YH4808 400 mg (repeat doses) — YH4808 400 mg (repeat doses)
  Arms: YH4808 400mg(repeat doses)
Drug: Placebo — 10 volunteers will be administered matched placebo.
  Other Names: 10 volunteers will be administered matched placebo.
  Arms: Placebo
Drug: Esomeprazole 40mg — 24 volunteers will be administered Esomeprazole 40mg
  Other Names: 24 volunteers will be administered Esomeprazole 40mg
  Arms: Esomeprazole 40mg

SUMMARY:
First in human study

DETAILED DESCRIPTION:
Study to evaluate the safety and tolerability, pharmacokinetics/pharmacodynamics (PK/PD) parameters of an escalating, single dose/repeat doses of YH4808 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers in the age between 20 to 45 years old
* Subjects who were determined to be appropriate through screening
* Weight: over 50kg, within ±20% of ideal body weight
* Subjects who signed written consent after receiving thorough explanation on trial purpose, content, and characteristics of investigational drug

Exclusion Criteria:

* Clinically significant disorder in liver, kidney, cardiovascular, respiratory system, endocrine system and CNS in the physical examination and clinical laboratory tests or a medical history of malignant tumor or psychological disease
* Medical history of gastrointestinal disease or acid restraining surgery, gastric/esophagus surgery (excluding appendectomy, hernia surgery)
* A history of hypersensitivity to drugs or clinically significant allergic disease
* Clinically significant abnormal values in blood chemistry(≥ 1.5 fold of normal upper limit in the levels of SGOT, SGPT)
* Subjects who were unable to be applicable for pH meter catheter
* Subjects who had a history of drug abuse or who had a positive results on urine drug screening
* Subjects who had taken usual dose of any prescription drugs within 14 days before the treatment or who had used usual dose of OTC drugs within 7 days before the treatment(cf, be able to be enrolled in this study according to an investigatory consideration)
* Subjects who participated in another clinical trial within 3 months before enrolling in this study
* Subjects who donated whole blood within 2 months or component blood within 1 month or who are donated within 1 month before the treatment
* Subjects who drank Over 21 units/week of alcohol or subjects who weren't able to stop drinking alcohol during the hospitalization
* Subjects who stopped smoking within 3 months before the treatment
* Subjects who had a beverage containing grapefruits within 24hrs before the hospitalization or who had a beverage containing grapefruits during the hospitalization
* Subjects who had a beverage containing caffeine during the hospitalization
* H.pylori positive results on the Urease breath test(Only repeat doses)
* Subjects with clinically significant observations considered as unsuitable based on medical judgment by investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the PKs, PDs, safety and tolerability of escalating, single/multiple oral doses of YH4808 | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Clinical trials center, Seoul national university hospital, Seoul, South Korea